CLINICAL TRIAL: NCT06416488
Title: The Effect of High-Intensity Interval Training(HIIT) on Cardio-metabolic Indicators in School-age Children With High Cardiovascular Diseases Risk--a Randomised Intervention Trial
Brief Title: High-Intensity Interval Training(HIIT) on Cardio-metabolic Risk in School-age Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-TABATA
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Syndrome, Metabolic
Keywords: Cardiovascular diseases; Metabolic disorders; High-Intensity Interval Training; School-aged children; Childhood obesity
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Metabolic Diseases; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT group (Experimental): HIIT group will follow modified HIIT in Tabata mode, at least 3 times per week, with 3-month compulsory period and 9-month follow-up period. General health education on promoting health diet and exercise will be sent to HIIT group via offline and online promotion materials during the whole study period of 12 months.
  Interventions: Behavioral: HIIT intervention; Behavioral: General health education
- General health education group (Active Comparator): General health education on promoting health diet and exercise will be sent to general health education group via offline and online promotion materials during the whole study period of 12 months.
  Interventions: Behavioral: General health education

INTERVENTIONS:
Behavioral: HIIT intervention — Modified HIIT in Tabata mode, which followed a pattern of 3 sets, with each set consisting of 4 repetitions of 20 seconds of high-intensity exercise followed by 10 seconds of rest, at least 3 times per week.
  Arms: HIIT group
Behavioral: General health education — General instructions on promoting healthy diet and exercise, primarily by sending offline and online promotion materials to participants.

SUMMARY:
This study aims to evaluate the health promotion effects of high-intensity interval training (HIIT) intervention on school-age children who are at high risk for cardiovascular disease (CVD), as well as the long-term adherence and acceptability of HIIT in this population for future application.

DETAILED DESCRIPTION:
Evidence shows that physical activity is positively associated with cardiovascular and metabolic health in children and adolescents, including promoting lipid health, regulating blood pressure levels, and glucose metabolism. Physical activity intervention for overweight or obese children can lower body mass index, total fat mass, and abdominal fat mass, and further prevent chronic diseases such as cardiovascular and metabolic diseases. High-intensity interval training (HIIT) has been a recent research focus. Previous studies have demonstrated that HIIT can contribute to improving body composition, reducing visceral fat, and enhancing cardiovascular and pulmonary function. Moreover, compared to other trainings, HIIT is time-efficient and adaptable to various sports, thus leading to higher compliance.

However, there has been a lack of evidence regarding the intervention effects of this exercise in overweight and obese children and adolescents, and whether it can impact or even reverse cardio-metabolic risks remains unknown.

Therefore, this intervention trial might have implications and practical significance on the feasibility of promoting HIIT among this population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-18 years at baseline.
* At least one of the following cardio-metabolic abnormalities:

  1. Prediabetes (Impaired fasting glucose: 5.6 ≤ fasting blood glucose level ≤ 6.9 mmol/L; or Impaired glucose tolerance: 7.8 ≤ blood glucose level after 2 hours postprandial ≤ 11.0 mmol/L).
  2. Lipid abnormalities (High-density lipoprotein cholesterol ≤ 1.04 mmol/L; or Low-density lipoprotein cholesterol ≥ 3.37 mmol/L; or Triglycerides ≥ 1.70 mmol/L, or Total cholesterol ≥ 5.18 mmol/L).
  3. Elevated blood pressure (Systolic/diastolic blood pressure consistently higher than the 90th percentile for gender, age, and height; or systolic/diastolic blood pressure ≥ 120/80 mmHg).
* Written consent from participants and their guardians.

Exclusion Criteria:

* Previously diagnosed with heart failure, severe malnutrition, immune deficiency, liver or kidney disease, cancer, or other diseases deemed unsuitable for participation.
* Taking weight loss drugs, or undergone weight loss surgery.
* Attending behavior-based intervention programs (exercise or diet) within a year.
* Regular HIIT (at least once per week).
* Secondary obesity, such as neuropsychiatric disorders, endocrine disorders, sleep apnea syndrome, or other conditions.
* Unable to take interventions due to health conditions, such as joint diseases, fractures, injuries.
* Other situations unsuitable for participation.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reversal of at least one cardio-metabolic abnormalities | 3rd month since baseline
  The primary outcome is a composite outcome that will be measured by combining multiple reverse outcomes of the following cardiometabolic abnormalities: (1) prediabetes; (2) lipid abnormalities; (3) elevated blood pressure. It is defined as occurring if any cardiometabolic abnormality has a reversal outcome at 3rd month of study phrase.
  Reversal of cardiometabolic abnormalities is defined as: at 3rd month of study phrase, at least one of the following status changed from abnormal at baseline to normal:
  i. Prediabetes; ii. Lipid abnormalities; iii. Elevated blood pressure.

SECONDARY OUTCOMES:
Number of participants with reversal of at least one cardio-metabolic abnormalities | 12th month since baseline
  It is a composite outcome that will be measured by combining multiple reverse outcomes of the following cardiometabolic abnormalities: (1) prediabetes; (2) lipid abnormalities; (3) elevated blood pressure. It is defined as occurring if any cardiometabolic abnormality has a reversal outcome at 12th month of study phrase.
  Reversal of cardiometabolic abnormalities is defined as: at 12th month of study phrase, at least one of the following status changed from abnormal at baseline to normal:
  i. Prediabetes; ii. Lipid abnormalities; iii. Elevated blood pressure.
Body mass index | 3rd and 12th month since baseline
  Body mass index(BMI) will be calculated by body weight(kg)/(height(m)^2), based on BMI z score and percentiles by sex and age according to Chinese children growth curves. Body weight and height will be measured by trained professionals.
Waist-to-height ratio | 3rd and 12th month since baseline
  Waist-to-height ratio(WHtR) will be calculated by waist circumference(cm)/height(cm). Waist circumference and height will be measured by trained professionals.
Body fat (%) | 3rd and 12th month since baseline
  Body fat(%) will be directly derived from non-invasive DEX body composition analyser, assessed by professional operator.
Resting metabolic rate | 3rd and 12th month since baseline
  Average amount of calories(kcal) when at complete rest (2 hours after meals), measured by a Parvo Medics TrueOne 2400 mask to measure exchanges of gases.
Maximal oxygen uptake（ml/min/kg) | 3rd and 12th month since baseline
  Maximal oxygen uptake(VO2max) will be measured by a Parvo Medics TrueOne 2400 mask after treadmill (Pulsar 4.0，h/p/Cosmos Sports and Medical GMBH , Germany).
Sleep quality | 3rd and 12th month since baseline
  Sleep quality monitoring for 1 week using sleep watch （Micro Motionlogger Watch）to measure total duration of sleeping (minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No